CLINICAL TRIAL: NCT01409187
Title: IPI-Biotherapy for Patients With Metastatic Melanoma Previously Treated With Cytotoxic Drugs
Brief Title: IPI-Biotherapy for Patients Previously Treated With Cytotoxic Drugs With Metastatic Melanoma
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0074
Record Dates: First submitted 2011-08-02; First posted 2011-08-04 (Estimated); Last update posted 2012-01-26 (Estimated); Status verified 2012-01

CONDITIONS: Melanoma
Keywords: Melanoma; Metastatic Melanoma; Cytotoxic Drugs; IPI-Biotherapy; Ipilimumab; Yervoy; BMS-734016; MDX010; Interferon; IFN Alpha-2b; Intron A; Interferon Apha-2b; Interleukin-2; IL-2; Aldesleukin; Proleukin
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab; Interferons; Introns; aldesleukin; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ipilimumab + Interferon + Interleukin-2 (Experimental): Ipilimumab starting dose 2 mg/kg intravenous (IV) day 1 only; IFN alfa-2b at 5 million U/m2 subcutaneously daily for 5 days starting day 1; IL-2 at 9 million IU/m^2 daily IV continuous infusion for 4 days on days 2-5.
  Interventions: Drug: Ipilimumab; Drug: Interferon; Drug: Interleukin-2 (Aldesleukin)

INTERVENTIONS:
Drug: Ipilimumab — Starting dose 2 mg/kg by vein on day 1 of each of the four 3-week cycles (Phase II is maximum tolerated dose (MTD) from Phase I). During Consolidation and Maintenance phases one dose every 12 weeks.
  Other Names: Yervoy; BMS-734016; MDX010
Drug: Interferon — 5 million U/m2 subcutaneously daily for 5 days starting day 1 of each Induction and Consolidation cycle.
  Other Names: IFN Alpha-2b; Intron A; Interferon Alpha-2b
Drug: Interleukin-2 (Aldesleukin) — 9 million IU/m^2 daily by vein by continuous infusion for 4 days (total of 96 hours, days 2-5) starting day 2 of each Induction and Consolidation cycle.
  Other Names: IL-2; Aldesleukin; Proleukin

SUMMARY:
The goal of the Phase I part of this clinical research study is to find the highest tolerable dose of the drug Yervoy (ipilimumab) that can be given with the drugs Intron-A (interferon alfa-2b) and Proleukin (aldesleukin, IL-2) to patients with metastatic melanoma. The safety of this combination will also be studied in Phase I. The goal of Phase II is to learn if this combination can help to control metastatic melanoma.

Ipilimumab, interferon alfa-2b, and aldesleukin are designed to block the activity of cells that decrease the immune system's ability to fight cancer.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a study group based on when you join this study. Up to 5 groups of 3-6 participants will be enrolled in the Phase I portion of the study, and up to 64 participants will be enrolled in Phase II.

If you are enrolled in the Phase I portion, the dose of ipilimumab you receive will depend on when you joined this study. The first group of participants will receive the lowest dose level of ipilimumab. Each new group will receive a higher dose of ipilimumab than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of ipilimumab is found.

If you are enrolled in the Phase II portion, you will receive ipilimumab at the highest dose that was tolerated in the Phase I portion.

All participants will receive the same dose level of interferon alfa-2b and aldesleukin.

Study Drug Administration:

The study drugs will be given in 3 stages: induction, consolidation, and maintenance.

Induction:

Induction will last 12 weeks. You will receive the study drugs in up to four 3-week cycles:

* You will receive ipilimumab by vein over 90 minutes on Day 1 of each cycle.
* You will receive aldesleukin in the hospital by vein as a continuous infusion on Days 2-5 of each cycle.
* You will receive interferon alfa-2b as an injection under your skin on Days 1-5 of each cycle.

Consolidation:

Consolidation will last 12 weeks. You will receive the study drugs in up to four 3-week cycles:

* You will receive ipilimumab by vein over 90 minutes on Day 1 of Cycle 1.
* You will receive aldesleukin in the hospital by vein as a continuous infusion on Days 2-5 of each cycle.
* You will receive interferon alfa-2b as an injection under your skin on Days 1-5 of each cycle.

Maintenance:

Maintenance will last about 1½ years. You will receive ipilimumab by vein over 90 minutes on Day 1 of up to six 12-week cycles.

Other Drugs:

You will be given other drugs to help lower the risk of side effects. The study staff will tell you about these drugs, how they will be given, and the possible risks.

Study Visits:

Before each cycle (+/- 3 days):

* You will be asked about any drugs you may be taking and any side effects you may have had.
* Your performance status will be recorded.
* Your vital signs will be measured.
* Blood (about 1 teaspoon) will be drawn for routine tests and tests of your liver and kidney function.
* If you are able to become pregnant, you will have a blood (about 1 teaspoon) or urine pregnancy test.

Every week, blood (about 1 teaspoon) will be drawn for routine tests.

At the end of each cycle, you will have a physical exam, including measurement of your weight. Any tumor that can be felt with the hands will be measured during the physical exam to see if it has changed size.

Every 2 cycles (+/- 7 days), you will have a chest x-ray and CT or MRI scans to check the status of the disease.

Anytime the doctor thinks it is needed, photos of the skin lesions will be taken. Your private areas will be covered (as much as possible), and a picture of your face will not be taken unless there are lesions on your face.

Length of Study:

You may continue taking the study drugs for up to 2 years. You will no longer be able to take the study drugs if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over once you have completed the end-of-treatment visit and follow-up.

End-of-Treatment Visit:

Within 14 days after you stop the study therapy, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your vital signs and weight.
* Your performance status will be recorded.
* You will be asked about any drugs you may be taking and any side effects you may have had.
* Blood (about 2 tablespoons) will be drawn for routine tests.
* If the doctor thinks it is needed, you will have a CT or MRI scan.

Every 2 months for up to 3 years, you will also be contacted by phone or during a clinic visit to see how you are doing.

This is an investigational study. Ipilimumab, interferon alfa-2b, and aldesleukin are FDA approved and commercially available to treat melanoma. Giving these drugs in combination is investigational.

Up to 88 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically documented diagnosis of advanced stage IV or unresectable stage III melanoma are eligible.
2. They should have recurrent melanoma with measurable or evaluable sites of disease, 1.0 cm or larger, in order to assess the response to treatment by the immune-related response criteria (irRC).
3. Phase I: Patients with prior therapy who do not have alternative treatment of higher priority will be eligible. Phase II: the patient may have been treated with cytotoxic drugs or targeted therapies but not with IL-2, interferon and anti-CTLA4 drugs for metastatic disease. Adjuvant ipilimumab will not be permitted. Only adjuvant interferon will be permitted. Prior radiation therapy for metastatic melanoma is permitted provided the patient has unirradiated metastatic sites for response evaluation and has fully recovered from its toxicity.
4. Patients between 18 years of age and 65 years of age with an ECOG performance status of 0, 1 or 2 will be eligible.
5. They should have normal blood counts with a white blood count (WBC) count of more than or equal to 3000/mm^3 an absolute neutrophil count of more than or equal to 1500/mm^3 and a platelet count of more than 100,000/mm^3 and have no impairment of renal function (serum creatinine less than 1.1 mg/dl for females and less than 1.4 mg/dl for males), hepatic function (serum bilirubin level of less than 1.2 mg/dl) and no evidence of significant cardiac or pulmonary dysfunction.
6. They should have no significant intercurrent illness such as an active infection associated with fever lasting more than 24 hours requiring antibiotics, uncontrolled psychiatric illness, hypercalcemia (calcium greater than 11 mg), or active gastrointestinal (GI) bleeding.
7. Females of child-bearing potential (non-childbearing is defined as greater than one year post-menopausal or surgically sterilized) must use acceptable contraceptive methods( abstinence, intrauterine device, oral contraceptive or double barrier devices) and must have a negative serum or urine pregnancy test within 14 days prior to beginning treatment on this trial. Sexually active men must also use acceptable contraceptive methods for the duration of time on study.

Exclusion Criteria:

1. Patients with bone metastases only.
2. Patients with brain metastases unless all of their metastatic brain lesions have been resected or treated with stereotactic radiotherapy with gamma rays and they are off corticosteroids. Patient should not have significant brain edema. Patients with spinal cord compression and leptomeningeal disease. No major surgery or radiation therapy within 21 days before starting treatment.
3. Patients with significant cardiac illness such as symptomatic coronary artery disease or previous history of myocardial infarction, impaired left ventricle function (Ejection Fraction less than 50%) on account of any organic disease such as hypertension or valvular heart disease or serious cardiac arrhythmia requiring therapy. Patients will be evaluated by the investigator or his designee.
4. Patients with significant impairment of pulmonary function on account of chronic bronchitis or chronic obstructive pulmonary disease (COPD) which has resulted in impairment of vital capacity of FEV1 to less than 65% of predicted normal values.
5. Patients with symptomatic effusions on account of pleural, pericardial or peritoneal metastases of melanoma.
6. Patients who are unable to return for follow-up visits as required by this study.
7. Patients with a history of second malignant tumor, other than the common skin cancers - basal and squamous carcinomas, within the past 3 years and uncertainty about the histological nature of the metastatic lesions. Cases with other types of malignancies should be reviewed and decided by the Principal Investigator (PI) of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-10; Primary Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Progression Free survival (PFS) | Assessed at 6-months then until disease progression or death.
  Progression-free survival determined from the start of the study until disease progression or death, whichever is first and estimated using the method of Kaplan-Meier.

CONTACTS AND LOCATIONS:
Overall Officials: Agop Y. Bedikian, MD,BS, Principal Investigator — UT MD Anderson Cancer Center

REFERENCES:
- See also: UT MD Anderson Website — http://www.mdanderson.org